CLINICAL TRIAL: NCT02758639
Title: Wonders & Worries: A Clinical Trial of a Psychosocial Intervention for Children Who Have a Parent With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Wonders & Worries (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201502573
Record Dates: First submitted 2016-04-25; First posted 2016-05-02 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Cancer; Psychological Adjustment
Keywords: parental cancer; children psychosocial adjustment; psychosocial intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- W & W Intervention (Experimental): Wonders & Worries Psychosocial intervention is a 6 week group or individual sessions for children who have a parent with cancer focusing on psycho-educational information about cancer, treatment and its side effects, feelings expression, positive coping strategies, and family communication about the illness.
  Interventions: Behavioral: Wonders & Worries Psychosocial Intervention
- Wait list control (Other): Wait list group will complete baseline, 6 week and 8 week follow up measures and then will be enrolled to receive W & W intervention.
  Interventions: Behavioral: Wonders & Worries Psychosocial Intervention

INTERVENTIONS:
Behavioral: Wonders & Worries Psychosocial Intervention — Session 1: Getting to Know Each Other The goal is to create a sense of safety within the group so that the children feel comfortable discussing difficult topics. Session 2: Cancer Education to provide developmentally appropriate education about the illness, treatment, and side effects. Session 3: Cancer Treatment Center Tour: This session consists of a treatment center tour and education about treatment plan involved in family's care in a safe environment. Session 4: Feelings: The focus of this session is expression and validation of all feelings the children may experience. Session 5: Stress and Coping: Goal is to emphasize the different ways individuals cope and differentiate positive vs. negative coping strategies. Session 6: Hopes for the Future/Closure: An emphasis is made on the idea that positive things may evolve from the most difficult circumstances.

SUMMARY:
Parental cancer can cause substantial behavioral and emotional distress in both parent and child. Parents struggle with talking with their child about their cancer and supporting the child during treatment. Over 73% of patients with children desire information and services to support their children yet only 9% of these families report receiving this support. The purpose of this study is to evaluate the Wonders & Worries psychosocial intervention designed for children ages 5-14 who have a parent diagnosed with early stage cancer.This study is a randomized controlled clinical trial (RCT) evaluating the Wonders & Worries group and individual intervention for school age children (5 -14 years old) who have a parent with cancer. Families will be enrolled at the time of initial parent consultation, given informed consent, and then randomized either to the intervention group of 30 families or the wait-listed control group of 30 families. Both groups will be given a series of standardized validated assessment instruments including the Revised Children's Manifest Anxiety Scale (RCMAS), the Child Behavior Checklist (CBCL), and the Family Communication Scale FACES IV at baseline, post intervention, and 8 week follow up. Upon completion of the follow up measures, families in the wait-listed control group will be enrolled into the intervention. Parent exit interviews for both groups will be used to measure parent-reported child outcomes and program utility.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the Wonders & Worries psychosocial intervention designed for children ages 5-14 who have a parent diagnosed with early stage cancer. The Wonders & Worries program curriculum is a psychosocial intervention that was designed to address the communication and distress issues raised in prior descriptive research and to respond to the limitations of current research. The goals of the program are to improve children's behavioral-emotional adjustment to their parent's cancer, improve parenting behavior (parenting quality, skills and self-efficacy), and increase family communication about the illness. The aim of the current study is to evaluate the efficacy of the Wonders & Worries program on child and parent outcomes within a randomized clinical trial.

Wonders & Worries is an Austin based non-profit agency. Wonders & Worries works with families in all stages of survivorship, who are affected by any serious or chronic physical illness.

The fully scripted intervention involves 6 group or individual sessions for the children, each of which is briefly summarized, in Table 1. Families will be enrolled at the time of initial parent consultation at Wonders & Worries, given informed consent, and then randomized either to the intervention group of 30 families or the wait-listed control group of 30 families. Both groups will be given a series of standardized validated assessment instruments including the Revised Children's Manifest Anxiety Scale (RCMAS), the Child Behavior Checklist (CBCL), the Family Communication Scale FACES IV, and the AMMI-EC3- About My Mommy's Illness at baseline, post intervention, and 8 week follow up. Upon completion of the follow up measures, families in the wait-listed control group will be enrolled into the intervention. Parent exit interviews for both groups will be used to measure parent-reported child outcomes and program utility.

The intervention will be provided by Wonders & Worries certified child life specialists. Child life specialists are professionals trained to help children and their families understand and manage challenging life events and stressful health care experiences. By using play, recreation, education, self-expression and theories of child development, these specialists help promote the psychological well-being and optimum development of children and families faced with stressful situations. At Wonders & Worries all services are provided by master's prepared certified child life specialists.

ELIGIBILITY:
Inclusion Criteria:

* Families with children ages 5-14 at time of study. Children have a parent with early stage cancer, and are English-speaking.

Exclusion Criteria:

* Children are not living in the home with the ill parent at least 50% of the time. Non-English speaking families.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2018-08-19 (Actual)

PRIMARY OUTCOMES:
Change in Child's Anxiety level (RCMAS) from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  Revised Children's Manifest Anxiety Scale - child self report
Change in Child's Emotional/Behavioral Status (CBCL) from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  Child Behavior Checklist - parent report
Change in Family Communication Scale FACES IV from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  parent & child report
Change in The Family Quality of Life Scale (FQOL) from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  parent & child report
Change in Cancer Self-Efficacy Scale (CASE) from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  parent report of parenting self efficacy
Change in Spielberger State-Trait Anxiety Inventory (STAI) from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  parent self report of anxiety
Change in Depression scale (CES-D) from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  parent self report of depression
Change in Parenting Concerns Questionnaire (PCQ) for adults with cancer from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  parent self report
Change in child's worries about their parent's illness from baseline to 6 weeks and 8 week follow up | Baseline, 6 week, 8 week follow up
  child self report of worries related to parent's illness AMMI-EC3- About My Mommy's Illness

CONTACTS AND LOCATIONS:
Overall Officials: Farya Phillips, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips F, Prezio EA. Wonders & Worries: evaluation of a child centered psychosocial intervention for families who have a parent/primary caregiver with cancer. Psychooncology. 2017 Jul;26(7):1006-1012. doi: 10.1002/pon.4120. Epub 2016 Mar 8. PMID 26954773
- [Derived] Phillips F, Prezio EA, Currin-McCulloch J, Jones BL. Wonders & Worries: A randomized clinical trial of a psychosocial intervention for children who have a parent with cancer. Psychooncology. 2022 Aug;31(8):1399-1411. doi: 10.1002/pon.5943. Epub 2022 Apr 29. PMID 35470518